CLINICAL TRIAL: NCT01542528
Title: Integrated Brain, Body and Social Intervention (IBBS) for Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Integrated Brain, Body and Social Intervention for Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: IBBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Hamden Public Schools, Connecticut (Unknown); C8Sciences (Industry); BeCaid China (Unknown); Peking University (Other); Capital Medical University (Other); Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11100009142; R01HD070821 (NIH)
Record Dates: First submitted 2012-02-23; First posted 2012-03-02 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; Executive function; Inhibitory control; Computer games; Sports activities; Good Behavior Game
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IBBS (Experimental): Combination of computer-presented brain exercises with a physical education curriculum designed to enhance sustained attention, inhibitory control and other executive capacities. Groups of 10 students incorporating the Good Behavior Game. Two-hour sessions four days a week: classroom with computers (45-60 mins) plus sports activities in the gymnasium (45-60 mins) extending over a total 15 weeks (60 sessions).
  Interventions: Behavioral: IBBS
- Treatment as Usual (TAU) (No Intervention): Whatever care arrangement the parents have arranged for their child during the same two hour period over the same 15 week period.

INTERVENTIONS:
Behavioral: IBBS — Combination of computer-presented brain exercises with a physical education curriculum designed to enhance sustained attention, inhibitory control and other executive capacities. Groups of 10 students incorporating the Good Behavior Game. Two-hour sessions four days a week: classroom with computers (45-60 mins) plus sports activities in the gymnasium (45-60 mins) extending over a total 15 weeks (60 sessions).
  Arms: IBBS

SUMMARY:
The investigators are conducting this randomized trial to determine if IBBS (Integrated Brain, Body, and Social)intervention is an effective treatment for ADHD (attention Deficit Hyperactivity Disorder) in two culturally distinct settings; Hamden and New Haven, Connecticut and Beijing, China. A subgroup of the children in the US will also participate in an EEG study before and after IBBS and will be compared to a group of typically developing children.

IBBS combines computer-presented brain exercises with a physical education curriculum, all of which is designed to be fun, as well as to enhance sustained attention, inhibitory control and other executive capacities.

IBBS is a school-based program in which groups children (composed of children with ADHD, children at risk for ADHD, and typically developing children) alternate between a classroom setting and the gymnasium four days a week for 15 weeks. These mixed age groups will be composed of children with ADHD, children at-risk for ADHD, and typically developing children. Although IBBS takes place in a group setting, the computer game component individualizes instruction to maximize benefit for each child.

During the last year of the grant, we will be introducing a pilot study of an organizational skills training (OST) that will provide individualized parent and child training for improved executive functioning in children randomized to the OST plus home-based program.

DETAILED DESCRIPTION:
Purpose Attention Deficit Hyperactivity Disorder (ADHD) is a neurodevelopmental disorder characterized by a failure to develop age-appropriate executive functions. Children with ADHD struggle to sustain and direct attention, to inhibit response to task-irrelevant stimuli and to contain and down regulate impulsive behavior. ADHD can interfere with healthy emotional and cognitive development. It often has a negative impact not only on a child's academic performance but also on peer and family relationships.

Medications are now widely used to treat ADHD in the US. However, we are evaluating another approach. Based on nearly 30-years of research by scientists at Yale and in China, our Integrated Brain, Body, and Social (IBBS) Intervention for ADHD combines computer-presented brain exercises with a physical education curriculum, all of which is designed to be fun, as well as to enhance sustained attention, inhibitory control and other executive capacities. Work by other investigators has also shown that computer exercises designed specifically to address aspects of neurocognitive dysfunction in ADHD can lead to improvements in working memory and sustained attention; however IBBS is the first intervention to combine advanced computer games with sports activities.

IBBS is a school-based program in which groups of 10 children (Kindergarten, First, and Second graders) alternate between a classroom setting (45 mins) and the gymnasium (45 mins) four days a week for 15 weeks. These mixed age groups will be composed of children with ADHD, children at-risk for ADHD, and typically developing children. Although IBBS takes place in a group setting, the computer game component individualizes instruction to maximize benefit for each child.

Since the social context has a clear impact on the expression of ADHD, we have also incorporated the "Good Behavior Game" (GBG) into these group activities. The GBG is intended to facilitate group participation and to enhance co-operative interactions both in the classroom and the gymnasium. The use of the GBG is another innovative feature of IBBS. Thus far, our preliminary results have shown that IBBS leads to a fundamental increase in cognitive abilities and focused attention.

We are conducting this randomized trial to determine if IBBS is an effective treatment for ADHD in two culturally distinct settings; Hamden, Connecticut and Beijing, China. A subgroup of the children in Hamden and New Haven will also participate in an EEG study before and after IBBS. Typically Developing Children will also be recruited from the community for the optional EEG study in order to ensure that the comparison group is well-matched with regard to age, gender, and intelligence quotient (IQ) to those children with ADHD who have already participated in the EEG study.

During the last year of the grant, we will be introducing a pilot study of an organizational skills training (OST) curriculum for parents and children. We ultimately aim to create a treatment for wide clinical application that can address primary pathology, promote more active and more complete neural development, and normalize developmental interactions with the environment. The treatment will be an aggressive early intervention at the time the relevant brain regions and systems are actively developing and clinical symptoms are first appearing.

We hypothesize in relation to clinical outcomes in the randomized controlled trial that:

1. Children receiving IBBS as after school program will show significantly greater improvement than children receiving treatment as usual in parent and teacher symptom ratings and laboratory tests of cognition.
2. Children's EEG data will be sensitive to the effects of IBBS.
3. Children receiving OST plus the home-based IBBS program will show significantly greater improvement than children receiving the home-based IBBS program alone.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls between 5 and 10 years of age, inclusive.
* Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV Diagnosis of ADHD (definite, probable, possible) based on a best estimate diagnosis using all available information.
* IQ of greater or equal to 80 on the Abbreviated IQ Test
* Currently not receiving any psychotropic medication or on a stable dose of medication prescribed for ADHD (psychostimulants, alpha agonists, atomoxetine, modafinil) for > 4 weeks.

Exclusion Criteria:

* English is a secondary language
* Current DSM-IV diagnosis requiring alternative treatment, e.g., Major Depression, Bipolar Disorder, Autism Spectrum Disorder, or a psychotic disorder.
* Presence of serious behavioral problems (tantrums, aggression, self-injury) for which another treatment is warranted or which could be too disruptive of the group treatment settings.
* Significant medical condition or injury identified by school personnel (that would normally identify these issues such as the school nurse, physical education teacher, or child's primary pediatrician) that would prohibit or limit the child's ability to perform the physical activity component of the IBBS (e.g. uncontrolled asthma or a musculoskeletal injury or condition.)
* Any restrictions that have been previously identified by the child's pediatrician to school personnel will, of course, be followed.
* Children with conditions normally prohibiting exercise will be excluded.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2012-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Leckman, MD, Principal Investigator — Yale University
Locations (5):
- United States (3):
  - Hamden Public Schools, Hamden, Connecticut
  - Department of Psychiatry, Yale University, New Haven, Connecticut
  - Yale Child Study Center, New Haven, Connecticut
- China (2):
  - Capital Medical University, Beijing, Beijing Municipality
  - Peking University, Beijing, Beijing Municipality

REFERENCES:
- [Background] Dovis S, Van der Oord S, Wiers RW, Prins PJ. Can motivation normalize working memory and task persistence in children with attention-deficit/hyperactivity disorder? The effects of money and computer-gaming. J Abnorm Child Psychol. 2012 Jul;40(5):669-81. doi: 10.1007/s10802-011-9601-8. PMID 22187093
- [Background] Embry DD. The Good Behavior Game: a best practice candidate as a universal behavioral vaccine. Clin Child Fam Psychol Rev. 2002 Dec;5(4):273-97. doi: 10.1023/a:1020977107086. PMID 12495270
- [Background] Fernandez A, Quintero J, Hornero R, Zuluaga P, Navas M, Gomez C, Escudero J, Garcia-Campos N, Biederman J, Ortiz T. Complexity analysis of spontaneous brain activity in attention-deficit/hyperactivity disorder: diagnostic implications. Biol Psychiatry. 2009 Apr 1;65(7):571-7. doi: 10.1016/j.biopsych.2008.10.046. Epub 2008 Dec 21. PMID 19103438
- [Background] Gaub M, Carlson CL. Behavioral characteristics of DSM-IV ADHD subtypes in a school-based population. J Abnorm Child Psychol. 1997 Apr;25(2):103-11. doi: 10.1023/a:1025775311259. PMID 9109027
- [Background] Ialongo NS, Werthamer L, Kellam SG, Brown CH, Wang S, Lin Y. Proximal impact of two first-grade preventive interventions on the early risk behaviors for later substance abuse, depression, and antisocial behavior. Am J Community Psychol. 1999 Oct;27(5):599-641. doi: 10.1023/A:1022137920532. PMID 10676542
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Klingberg T, Fernell E, Olesen PJ, Johnson M, Gustafsson P, Dahlstrom K, Gillberg CG, Forssberg H, Westerberg H. Computerized training of working memory in children with ADHD--a randomized, controlled trial. J Am Acad Child Adolesc Psychiatry. 2005 Feb;44(2):177-86. doi: 10.1097/00004583-200502000-00010. PMID 15689731
- [Background] Leckman JF, Sholomskas D, Thompson WD, Belanger A, Weissman MM. Best estimate of lifetime psychiatric diagnosis: a methodological study. Arch Gen Psychiatry. 1982 Aug;39(8):879-83. doi: 10.1001/archpsyc.1982.04290080001001. PMID 7103676
- [Background] MTA Cooperative Group. National Institute of Mental Health Multimodal Treatment Study of ADHD follow-up: changes in effectiveness and growth after the end of treatment. Pediatrics. 2004 Apr;113(4):762-9. doi: 10.1542/peds.113.4.762. PMID 15060225
- [Background] MTA Cooperative Group. National Institute of Mental Health Multimodal Treatment Study of ADHD follow-up: 24-month outcomes of treatment strategies for attention-deficit/hyperactivity disorder. Pediatrics. 2004 Apr;113(4):754-61. doi: 10.1542/peds.113.4.754. PMID 15060224
- [Background] Northup J, Broussard C, Jones K, George T, Vollmer TR, Herring M. The differential effects of teacher and peer attention on the disruptive classroom behavior of three children with a diagnosis of attention deficit hyperactivity disorder. J Appl Behav Anal. 1995 Summer;28(2):227-8. doi: 10.1901/jaba.1995.28-227. PMID 7601806
- [Background] Raggio DJ, Scattone D, May W. Relationship of the Kaufman Brief Intelligence Test-Second Edition and the Wechsler Abbreviated Scale of Intelligence in children referred for ADHD. Psychol Rep. 2010 Apr;106(2):513-8. doi: 10.2466/pr0.106.2.513-518. PMID 20524553
- [Background] Robbins TW. Shifting and stopping: fronto-striatal substrates, neurochemical modulation and clinical implications. Philos Trans R Soc Lond B Biol Sci. 2007 May 29;362(1481):917-32. doi: 10.1098/rstb.2007.2097. PMID 17412678
- [Background] Shalev L, Tsal Y, Mevorach C. Computerized progressive attentional training (CPAT) program: effective direct intervention for children with ADHD. Child Neuropsychol. 2007 Jul;13(4):382-8. doi: 10.1080/09297040600770787. PMID 17564853
- [Background] Shaw P, Sharp WS, Morrison M, Eckstrand K, Greenstein DK, Clasen LS, Evans AC, Rapoport JL. Psychostimulant treatment and the developing cortex in attention deficit hyperactivity disorder. Am J Psychiatry. 2009 Jan;166(1):58-63. doi: 10.1176/appi.ajp.2008.08050781. Epub 2008 Sep 15. PMID 18794206
- [Background] Swanson J, Lerner M, March J, Gresham FM. Assessment and intervention for attention-deficit/hyperactivity disorder in the schools. Lessons from the MTA study. Pediatr Clin North Am. 1999 Oct;46(5):993-1009. doi: 10.1016/s0031-3955(05)70168-1. PMID 10570701
- [Background] van Lier PA, Muthen BO, van der Sar RM, Crijnen AA. Preventing disruptive behavior in elementary schoolchildren: impact of a universal classroom-based intervention. J Consult Clin Psychol. 2004 Jun;72(3):467-78. doi: 10.1037/0022-006X.72.3.467. PMID 15279530
- [Background] Wexler BE, Anderson M, Fulbright RK, Gore JC. Preliminary evidence of improved verbal working memory performance and normalization of task-related frontal lobe activation in schizophrenia following cognitive exercises. Am J Psychiatry. 2000 Oct;157(10):1694-7. doi: 10.1176/appi.ajp.157.10.1694. PMID 11007730
- [Background] Bikic A, Christensen TO, Leckman JF, Bilenberg N, Dalsgaard S. A double-blind randomized pilot trial comparing computerized cognitive exercises to Tetris in adolescents with attention-deficit/hyperactivity disorder. Nord J Psychiatry. 2017 Aug;71(6):455-464. doi: 10.1080/08039488.2017.1328070. Epub 2017 Jun 9. PMID 28598701
- [Background] Li F, Zheng Y, Smith SD, Shic F, Moore CC, Zheng X, Qi Y, Liu Z, Leckman JF. A preliminary study of movement intensity during a Go/No-Go task and its association with ADHD outcomes and symptom severity. Child Adolesc Psychiatry Ment Health. 2016 Dec 12;10:47. doi: 10.1186/s13034-016-0135-2. eCollection 2016. PMID 27999615
- [Background] Kennedy D. Performance on a computerized cognitive remediation of students with attention deficit hyperactivity disorder. A thesis submitted to Yale School of Medicine in partial fulfillment of the requirements for the degree of doctor of medicine. January, 2013.
- [Result] Smith SD, Vitulano LA, Katsovich L, Li S, Moore C, Li F, Grantz H, Zheng X, Eicher V, Aktan Guloksuz S, Zheng Y, Dong J, Sukhodolsky DG, Leckman JF. A Randomized Controlled Trial of an Integrated Brain, Body, and Social Intervention for Children With ADHD. J Atten Disord. 2020 Mar;24(5):780-794. doi: 10.1177/1087054716647490. Epub 2016 May 13. PMID 27178060
- See also: website for company developing the computer programs to enhance cognitive development — http://www.c8sciences.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IBBS | Treatment as Usual (TAU)
Started | 61 | 56
Completed | 49 | 49
Not Completed | 12 | 7
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IBBS | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 59 | 54 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.6 (1.14) | 7.3 (1.17) | 7.4 (1.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 42 | 38 | 80
Race/Ethnicity, Customized [Number; unit: participants]
  White | 23 | 18 | 41
  African American | 11 | 11 | 22
  Hispanic | 7 | 8 | 15
  Asian | 12 | 9 | 21
  More than one race, other | 6 | 7 | 13
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 45 | 93
  China | 11 | 9 | 20
Clinician Rated SNAP Swanson, Nolan, and Pelham Rating Scale score [Mean (Standard Deviation); unit: units on a scale] — ADHD severity was measured by the Swanson, Nolan, and Pelham Rating Scale (SNAP)-IV-ADHD consists of 18 items that closely parallel in wording the diagnostic symptoms for ADHD as they appear in the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV. The range of scores are from 0 to 54. Higher scores indicate greater ADHD severity . The blinded assessors (Clinicians) used clinical judgement to provide an overall rating, based on all available information from the parents, teachers, and the assessors' own direct interactions with the child on the day of the assessment.
  units on a scale | 30.8 (7.9) | 29.9 (6.8) | 30.3 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in ADHD Severity From Baseline to End of Intervention
Description: ADHD severity was measured by the Swanson, Nolan, and Pelham Rating Scale (SNAP)-IV-ADHD consists of 18 items that closely parallel in wording the diagnostic symptoms for ADHD as they appear in the DSM-IV. The range of scores are from 0 to 54. Higher scores indicate greater ADHD severity . The blinded assessors (Clinicians) used clinical judgement to provide an overall rating, based on all available information from the parents, teachers, and the assessors' own direct interactions with the child on the day of the assessment.
Time Frame: End of intervention is at a maximum of 15 weeks from baseline.
Population: The analysis population are those with matched cases at 15 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IBBS | Treatment as Usual (TAU)
Number analyzed (Participants) | 51 | 47
units on a scale | 3.0 (6.56) | 3.2 (8.02)

2. Secondary Outcome: Overall Improvement
Description: Clinical Global Improvement Scale (CGI-I) - responders vs. non-responders. CGI is a seven point scale with the following anchor point: 1=Very Much Improved, 2=Much Improved, 3=Improved, 4=No change, 5=Minimally worse, 6=Much worse, 7=Very much worse. Participants with a score of 1, 2, or 3 at Endpoint were considered Responders; all others were considered non-responders.
Time Frame: 15 weeks for a total of 60 IBBS sessions vs. treatment as usual (TAU)
Population: The analysis population are those with matched cases at 15 weeks.
Measure: Number; unit: Percentage of participants
Arm/Group | IBBS | Treatment as Usual (TAU)
Number analyzed (Participants) | 51 | 47
Percentage of participants | 60.8 | 59.6

ADVERSE EVENTS:
Arm/Group | IBBS | Treatment as Usual (TAU)
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/54
Other Adverse Events (participants affected / at risk) | 13/59 | 0/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBBS (N=59) | Treatment as Usual (TAU) (N=54)
Minor incidents (scratches, bumped knees, etc) (Skin and subcutaneous tissue disorders) | 8 (10) | 0 (0)
Disruptive behaviors (Social circumstances) | 5 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No